CLINICAL TRIAL: NCT07041853
Title: The Effects of KSM-66 Ashwagandha (Withania Somnifera) Supplementation on Recovery and Muscle Strength in Academy Athletes
Brief Title: The Effects of KSM-66 Ashwagandha Supplementation on Recovery and Muscle Strength in Academy Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ramon Llull (Other)
Responsible Party: Principal Investigator, Blanca Roman-Viñas, MD, Professor, University Ramon Llull
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 05-03-2025
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Recovery; Strength; Exercise Training
Keywords: ashwagandha; athlete; recovery; performance; cortisol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KSM-66 Ashwagandha (Experimental): 600mg root extract KSM-66 Ashwagandha, once daily taken with dinner
  Interventions: Dietary Supplement: KSM-66 Ashwagandha
- Placebo (Placebo Comparator): 600mg organic chickpea flour, once daily taken with dinner
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: KSM-66 Ashwagandha — Root extract ashwagandha, KSM-66
  Arms: KSM-66 Ashwagandha
Dietary Supplement: Placebo — Organic chickpea flour
  Arms: Placebo

SUMMARY:
This double-blind, randomised, placebo-controlled trial will examine the effects of 42-day root extract ashwagandha (KSM-66) supplementation on recovery and muscle strength in male and female rugby and water polo players. Participants will receive either 600 mg of ashwagandha or a placebo daily. Outcomes include hormonal stress markers, perceived exertion, wellness, muscle soreness and strength and performance metrics (grip strength, jump tests, 1RM lifts, Bronco test).

DETAILED DESCRIPTION:
This double-blind, randomised, placebo-controlled trial aims to investigate the effects of ashwagandha (ASH) supplementation on recovery and muscle strength in male and female rugby and water polo players. Participants will supplement either KSM-66 ashwagandha (600 mg, standardised to 5% withanolides) or a placebo once daily for 42 days. The study will evaluate outcomes related to hormonal stress markers, perceived exertion, wellness, muscle soreness, and physical performance.

Primary biomarkers include cortisol, DHEA-S, testosterone, melatonin, alpha-amylase, and cortisone, assessed through saliva samples. Subjective measures will include the Borg Rate of Perceived Exertion Scale and the Hooper Index for sleep quality, stress, fatigue, and delayed onset muscle soreness (DOMS). Physical performance will be assessed using grip strength (CAMRY dynamometer), vertical jump tests (countermovement jump, squat jump), broad jump, 1-repetition maximum (1RM) tests for deadlift, bench press, and pull-up, as well as the Bronco test. Supplement satisfaction will be evaluated via questionnaire.

Participants' dietary intake will be recorded using a self-tracking method (Snap-N-Send) and analysed using Nutritics software; food diaries will serve as covariates in the final analysis. The study will be conducted in partnership with CN Poble Nou, a professional sports club in Barcelona, Spain.

Ashwagandha use is increasingly common among athletes despite limited evidence on appropriate dosing and performance outcomes. This study will contribute to scientific understanding of its potential short-term benefits, particularly in high-contact sports where managing cortisol and recovery is critical.

All participants will provide informed consent, and ethical considerations focus on safety, data privacy, and the right to withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18
* Healthy and free of disease
* Assigned as an athlete at CN Poble Nou sports academy

Exclusion Criteria:

* Allergies to nightshades such as tomato, aubergine, potatoes and peppers
* Active supplementation with other ergogenic aids (to not interfere with existing treatment)
* Medication or contraceptives (to not interfere with existing treatment)
* Liver conditions (to not interfere with existing treatment)
* Thyroid conditions (to not interfere with existing treatment)
* Diabetes or certain autoimmune conditions (to not interfere with existing treatment)
* Active pregnancy (to not interfere with existing treatment)
* No signing of the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Cortisol | Baseline and final measurement at 6 weeks
  Salivary cortisol
Hand grip | Baseline and final measurement at 6 weeks
  Hand grip strength in kilograms, CAMRY dynanometer

SECONDARY OUTCOMES:
Testosterone | Baseline and final measurement at 6 weeks
  Salivary testosterone
Melatonin | Baseline and final measurement at 6 weeks
  Salivary melatonin
DHEA-s | Baseline and final measurement at 6 weeks
  Salivary DHEA-s
Alpha-amylase | Baseline and final measurement at 6 weeks
  Salivary alpha-amylase
Cortisone | Baseline and final measurement at 6 weeks
  Salivary cortisone
Bronco test | Baseline and final measurement at 6 weeks
  Aerobic fitness test in minutes and seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Club Natació Poble Nou, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available upon reasonable request for academic research purposes.
Supporting Information: ICF

REFERENCES:
- [Derived] Coope OC, Otaegui E, Suarez M, Levington A, Abad-Sangra M, Lloyd B, Spurr TJ, Roman-Vinas B. Ashwagandha Root Extract Stabilises Physiological Stress Responses in Male and Female Team Sports Athletes During Pre-Season Training. Nutrients. 2026 Jan 12;18(2):230. doi: 10.3390/nu18020230. PMID 41599843